CLINICAL TRIAL: NCT06301737
Title: Effect of Stellate Ganglion Lidocaine Injection on Post-Stroke Pharyngeal Dysphagia
Brief Title: Lidocaine Injection: A Nove Block Therapy for Stroke-related Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad (Other)
Responsible Party: Sponsor-Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Organization: Ahmadu Bello University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-YanD
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Injections; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comprehensive rehabilitation+stellate ganglion block (Experimental): Patients enrolled are firstly numbered for privacy with software and divided into the observation group and the control group with. Additionally, the staffs involved in assessment would not participate in the intervention of the study. The treatment lasts 10 days.
  Interventions: Behavioral: Comprehensive rehabilitation; Drug: Lidocaine Hydrochloride
- comprehensive rehabilitation+placebo (Placebo Comparator): Patients enrolled are firstly numbered for privacy with software and divided into the observation group and the control group with. Additionally, the staffs involved in assessment would not participate in the intervention of the study. The treatment lasts 10 days.
  Interventions: Behavioral: Comprehensive rehabilitation; Procedure: Injection

INTERVENTIONS:
Behavioral: Comprehensive rehabilitation — All the participants are provided with the comprehensive rehabilitation (routine rehabilitation and swallowing function training). The routine rehabilitation included intervention for risk factors (blood pressure, blood lipids, blood glucose, smoking and alcohol restriction, exercise, etc.).
  Regrading swallowing function training, both groups are given swallowing function training, including 1) exercises of closure of the vocal folds, pharyngeal, and laryngeal muscles exercises, and respiratory muscle strength training, for 15 min each time and twice per day. 2) isotonic／isometric swallowing exercises, supraglottic swallowing exercises, for 20 min each time and twice per day. 3) effortful swallowing exercises, and cough reflex training, for 10 min each time and twice per day.
Procedure: Injection — the patients were provided with Injection. The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: comprehensive rehabilitation+placebo
Drug: Lidocaine Hydrochloride — the patients were provided with Stellate ganglion block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Other Names: Lidocaine
  Arms: comprehensive rehabilitation+stellate ganglion block

SUMMARY:
This was a multicenter randomized controlled study. 66 post-stroke patients with pharyngeal dysphagia were randomly allocated to the observation group (n=33) or the control group (n=33). Both groups were provided with comprehensive rehabilitation including routine rehabilitation and swallowing function training. Besides, the observation group additionally underwent the stellate ganglion block (SGB). At admission and after 20-day treatment, Kubota water swallowing test, video fluoroscopic swallowing study (VFSS), and Rosenbek penetration-aspiration scale (PAS) were used to assess swallowing function.

DETAILED DESCRIPTION:
Dysphagia is a frequent and potentially serious complication of stroke. However, there is no effective measure for the treatment of pharyngeal dysphagia in stroke patients. This study aims to explore the efficacy of stellate ganglion block in post-stroke pharyngeal dysphagic patients who received comprehensive rehabilitation. This was a multicenter randomized controlled study. 66 post-stroke patients with pharyngeal dysphagia were randomly allocated to the observation group (n=33) or the control group (n=33). Both groups were provided with comprehensive rehabilitation including routine rehabilitation and swallowing function training. Besides, the observation group additionally underwent the stellate ganglion block (SGB). At admission and after 20-day treatment, Kubota water swallowing test, video fluoroscopic swallowing study (VFSS), and Rosenbek penetration-aspiration scale (PAS) were used to assess swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ischemic stroke according to the diagnostic criteria, with the stroke occurring in the medulla oblongata and diagnosed as bulbar palsy.
* Upper Esophageal Sphincter did not open or opened ineffectively, with food residue or aspiration, revealed by Videofluoroscopic Swallow Study.
* Age >18 years.
* First-time stroke.
* Steady vital signs,
* Transferred or admitted to the Department of Rehabilitation Medicine within 15d after onset.

Exclusion Criteria:

* Allergy to Lidocaine injection or vitamin B12 injection;
* Severe cognitive impairment;
* Coagulation disorders;
* Severe dysfunction of organs including heart, lungs, kidney, liver, etc.;
* Complicated with other neurological diseases;
* Dysphagia caused by other diseases or reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Video fluoroscopic swallowing study | day 1 and day 10
  The patient was required to take a sitting position with the head naturally upright. Under the guidance of the examiner, the patient first swallowed 5ml of iohexol solution (50ml:17.5g in iodine terms). If the patient exhibited aspiration, the test would stop. If not, the patient was instructed to swallow 10ml of iohexol solution mixed with breadcrumbs, and the patient's swallowing condition was observed with immediate measures ready to take for safety. Specially, the esophageal phase was not included in the study, because it was commonly regarded as an independent phase. The swallowing were divided into 3 phases in this assessment: Oral phase, Pharyngeal phase, and Aspiration, with maximum 3,3,4 points were given to each phase. The total score was calculated as the final result. The final score was positively correlated with the swallowing function.

SECONDARY OUTCOMES:
Rosenbek penetration-aspiration scale | day 1 and day 10
  Based on VFSS, this assessment evaluated the patient's swallowing of contrast medium and whether there was retention, penetration, and aspiration. It included multiple items, each with the corresponding criteria, Specifically, whether the swallowed material entered the airway, passed through or contacted the vocal cords, and whether the patient exhibited the corresponding ability to clear. There were 8 levels in the results, with higher levels indicating more severe aspiration.
Functional Oral Intake Scale | day 1 and day 10
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The Functional Oral Intake Scale assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability. In general, the result below level 6 indicates unsafe for oral intake while level 6 and above indicates that eating via mouth can be safely conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group
Locations (1):
- Zhen No.1 Hos., Taiwan, China

IPD SHARING:
Plan to Share IPD: No